CLINICAL TRIAL: NCT00859677
Title: Immunologic Predisposition of HIV Patients to Develop Methicillin-Resistant Staphylococcus Aureus (MRSA) Colonization and Infection
Acronym: MRSA-2
Status: Completed | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Infectious Diseases Clinical Research Program (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IDCRP -023
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: HIV Infections; Staphylococcal Infections
Keywords: HIV; Methicillin-resistant Staphylococcus aureus (MRSA); HIV and Staphylococcus aureus infection
MeSH Terms: conditions — HIV Infections; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skin biopsy will be obtained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- 1: HIV-positive and MRSA negative
- 2: HIV-positive and MRSA infected (skin/soft tissue)
- 3: HIV-positive and MRSA colonized
- 4: HIV-negative and MRSA negative
- 5: HIV-negative and MRSA infected (skin/soft tissue)
- 6: HIV-negative and MRSA colonized

SUMMARY:
The purpose of this study is to investigate the role of T helper 17 cells (Th17) in the pathogenesis of MRSA infections.

ELIGIBILITY:
All participant inclusion criteria:

* Greater or equal to 18 years of age
* Willingness to undergo blood draw. Skin biopsy will be requested, but is optional

-AND-

HIV-positive and MRSA-negative Group:

* Documented positive HIV test result
* Negative colonization swabs for S. aureus within 14 days of enrollment
* No evidence of skin/soft tissue infection

HIV-positive and MRSA-Colonization Group:

* Documented positive HIV test result
* History of of colonization with MRSA w/in 14 days of study enrollment

HIV-positive and MRSA Infection Group:

* Documented positive HIV test result
* Skin/soft tissue infection with a positive wound culture showing MRSA within 7 days of enrollment
* MRSA infection is not associated with an intravenous catheter or other nosocomial procedure

HIV Negative groups:

* Same criteria used for the HIV-negative groups as listed above.
* No history of HIV infection.
* Willing to undergo an HIV blood test, which must have a negative result.

Exclusion Criteria:

* Women with positive urine pregnancy test within 7 days of study enrollment
* Women who are within 6 months of being postpartum or who are currently breastfeeding
* Subjects unable or unwilling to complete questionnaires and blood draw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-positive and negative patients with a recent screen for MRSA colonization or a history of MRSA infection will be asked to participate. Participants will be recruited by providers within the infectious disease clinics at the sites. In addtion, MRSA isolates will be monitored at the central laboratory and providers of patients with MRSA will be notified and asked to notify their patients of the opportunity to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-03; Primary Completion 2010-11 (Actual); Study Completion 2016-08-26 (Actual)

PRIMARY OUTCOMES:
To compare distribution of Th17 cells and their functionality, in the peripheral blood of HIV-positive patients who are infected with MRSA with that of HIV-positive patients who are not colonized or infected with Staphylococcus aureus. | 1 year

SECONDARY OUTCOMES:
Compare distribution of Th17 cells in the peripheral blood of groups of HIV-positive and HIV-negative participants who are colonized with MRSA as well as those who have a MRSA infection. | 1 year
Examine distribution of T cells, B cells, macrophages, dendritic cells, neutrophils, defensins, and IL-17 in T cell subsets in the skin | 1 year
Compare Th17 cells in peripheral blood of HIV-negative participants with MRSA infection with that of HIV-negative subjects not colonized of infected with Staph aureus. | 1 year
Collect information on factors that may play a role in development of MRSA colonization/infection. Includes demographic, hygienic, exercise-related, and sexual factors which may contribute to MRSA. | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland

REFERENCES:
- [Result] Utay NS, Roque A, Timmer JK, Morcock DR, DeLeage C, Somasunderam A, Weintrob AC, Agan BK, Estes JD, Crum-Cianflone NF, Douek DC. MRSA Infections in HIV-Infected People Are Associated with Decreased MRSA-Specific Th1 Immunity. PLoS Pathog. 2016 Apr 19;12(4):e1005580. doi: 10.1371/journal.ppat.1005580. eCollection 2016 Apr. PMID 27093273